CLINICAL TRIAL: NCT06181162
Title: YoPA - A Youth-centred Participatory Action Approach Towards Co-created Implementation of Socially and Physically Activating Environmental Interventions in Africa and Europe.
Brief Title: YoPA - A Youth-centred Participatory Action
Acronym: YoPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting Alexander (the Netherlands) (Unknown); Syddansk Universitet, Denmark (Unknown); Aalborg Municipality (Other); University of the Witwatersrand Johannesburg (South Africa) (Unknown); WITS Health Consortium (South Africa) (Unknown); Redeemer's University (Nigeria) (Unknown); Value Re-Orientation for Community Enhancement (Nigeria) (Unknown); Instituut voor Tropische Geneeskunde, Belgium (Unknown); COFAC Cooperativa de Formacao e Animacao Cultural CRL (Portugal) (Unknown); EMMA Communicatie B.V. (Unknown)
Responsible Party: Principal Investigator, Mai J M Chin A Paw, PhD, Prof.Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HORIZON Europe 101095423; 101095423 (Other Grant/Funding Number: EU HORIZON-HLTH-2022-DISEASE-07-03)
Record Dates: First submitted 2023-11-20; First posted 2023-12-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Health Promotion; Sleep; Screen Use
Keywords: Participatory Action Research; Health Promotion; Systems Approach; Adolescents; 24-hour movement behaviour; Physical activity; Urban health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: YoPA introduces teen-centred, evidence-informed co-creation to tackle the complex real-world challenge of unhealthy lifestyles and health inequalities. In urban environments in 'Minority World' countries (i.e., Denmark, the Netherlands) and 'Majority World' countries (i.e., Nigeria, South Africa), academic researchers will engage adolescents and other key stakeholders in local co-creation communities. Together with academic researchers and local stakeholders, adolescents will be central in 1) mapping the local system, including needs and opportunities; 2) tailoring interventions to the local context; 3) implementing, and 4) evaluating interventions guided by our novel SUPER-AIM framework assessing local Systems, User perspective, Participatory co-creation process, Reach, Effects, Adoption, Implementation, and Maintenance of interventions in an integrated manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents growing up in vulnerable life situations in four diverse urban environments. (Experimental)
  Interventions: Other: Social and/or physical environmental interventions

INTERVENTIONS:
Other: Social and/or physical environmental interventions — To be determined in the co-creation groups at the four sites (Denmark, the Netherlands, Nigeria, South Africa)

SUMMARY:
Background

A vast majority of adolescents do not meet guidelines for healthy physical activity, sedentary behaviour, and sleep, posing major risks for developing multiple non-communicable diseases. Unhealthy lifestyles seem more prevalent in urban than rural areas, with the neighbourhood environment as a mediating pathway linking urban living and poor health. How to develop and implement sustainable and effective interventions focused on adolescent health and wellbeing in urban vulnerable life situations is a key challenge and research gap. This paper describes the protocol of a Youth-centred Participatory Action (YoPA) project aiming to tailor, implement, and evaluate social and physical environmental interventions using an evidence-informed youth-centred co-creation approach, for structural improvement of the lifestyles of adolescents in urban vulnerable life situations.

Methods

In diverse urban environments in Denmark, the Netherlands, Nigeria, and South Africa, academic researchers will engage adolescents (12-19 years) growing up in vulnerable life situations and other key stakeholders (e.g., policy makers, urban planners, community leaders) in local co-creation communities. Together with academic researchers and local stakeholders, adolescents will take a leading role in mapping the local system for needs and opportunities; tailoring interventions to their local context; implementing and evaluating interventions during participatory meetings over the course of three years. YoPA applies a participatory mixed methods design guided by the newly developed SUPER-AIM framework assessing: (i) the local Systems, (ii) User perspectives, (iii) the Participatory co-creation process, (ii) Effects, iv) Reach, (vi) Adoption, (vii) Implementation, and (viii) Maintenance of interventions, in an integrated manner.

Discussion

YoPA aims to fill various research gaps, including the development of a practical protocol guiding the application of co-creation to tailor evidence-informed interventions to divers, multi-country contexts. Additionally, it focuses on advancing the research gap in physical activity and health within Sub-Saharan Africa and the involvement of adolescents in shaping their physical and social environments. Academic researchers envision that the YoPA co-creation approach will serve as a guide for participation of adolescents in vulnerable life situations in implementation of health promotion and urban planning in Europe, Africa and globally.

ELIGIBILITY:
Inclusion Criteria:

* aged 12 to 18 years
* living in a disadvantaged area in Aalborg (Denmark), Amsterdam (the Netherlands), Osogbo (Nigeria), or Soweto (South Africa)
* active informed consent by the adolescents and at least one parent/caregiver where applicable for the participation of the adolescent

Exclusion Criteria:

* none

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
24-h movement behaviours (i.e., physical activity, sedentary behaviour and sleep). | Pre-implementation, directly after implementation, and 3-6 months after implementation of the intervention.
  24-h movement behaviours will be assesed by questionnaire and accelerometers.
  The questionnaire contains questions on sleep (time spent on sleeping on a school day and weekend day, number of days feeling sleepy in the last week), physical activity (time spent in physical activity) and screentime (watching a screen on weekdays and weekend days).
Physical activity and associated environmental characteristics in selected outdoor spaces | Pre-implementation, directly after implementation, and 3-6 months after implementation of the intervention.
  SOPLAY is a validated tool for directly observing physical activity and associated environmental characteristics in free play settings (e.g., recess and lunch at school). SOPLAY provides objective data on the number of participants and their physical activity levels during play and leisure opportunities in targeted areas. Separate scans are made for males and females, and simultaneous entries for contextual characteristics of areas including their accessibility, usability, and whether or not supervision, organized activities, and equipment are provided. The predominant type of activity engaged in by area users is also recorded (e.g., basketball, dance).

SECONDARY OUTCOMES:
Agency | Pre-implementation, directly after implementation, and 3-6 months after implementation of the intervention.
  Agency is assessed by two domains scales of the Global Early Adolescent Study (GEAS): voice and freedom of movement, The voice scale conists of seven items. the freedom of movement scale consists of six items. Each item is scored from 0 (never / rarely) to 2 (often), and each domain is scored as the mean of the items scores. Higher domain scores indicate a higher level of voice and freedom of movement.
Wellbeing | Pre-implementation, directly after implementation, and 3-6 months after implementation of the intervention.
  Wellbeing is assessed by the PROMIS short form 8b Pediatric Life Satisfaction. This short form Pediatric Life Satisfaction consists of 8 items, which are scored from 1 (never) to 5 (almost always). Total scores are calculated by applying the original U.S. IRT model to the data and estimating the level of functioning of the patient (θ). This level of functioning is transformed into a T-score and is calculated by the formula (θ × 10) + 50, with higher scores representing higher levels of life satisfaction.
Peer relationships | Pre-implementation, directly after implementation, and 3-6 months after implementation of the intervention.
  Peer relationships is assessed by the PROMIS short form 8a Pediatric Peer Relationships. The Pediatric Peer Relationships short form consists of 8 items, which are scored from 1 (never) to 5 (almost always). Total scores are calculated by applying the original U.S. IRT model to the data and estimating the level of functioning of the patient (θ). This level of functioning is transformed into a T-score and is calculated by the formula (θ × 10) + 50, with higher scores representing higher levels of peer relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Mai JM Chin A Paw, Prof.Dr., Principal Investigator — Amsterdam UMC, location VUmc; Teatske M Altenburg, A/Prof.Dr., Principal Investigator — Amsterdam UMC, location VUmc; Jasper Schipperijn, Prof.Dr., Principal Investigator — Syddansk Universitet; Charlotte S Pawlowski, A/Prof.Dr., Principal Investigator — Syddansk Universitet; Adewale L Oyeyemi, A/Prof.Dr., Principal Investigator — Arizona State University; Bruno Marchal, Prof.Dr., Principal Investigator — Instituut voor Tropische Geneeskunde; António L Palmeira, A/Prof.Dr., Principal Investigator — COFAC Cooperativa de Formacao e Animacao Cultural CRL; Marlene Nunes Silva, A/Prof.Dr., Principal Investigator — COFAC Cooperativa de Formacao e Animacao Cultural CRL; Dayo Omotoso, Dr., Principal Investigator — Redeemer's University; Lisa Ware, Dr., Principal Investigator — University of Witwatersrand, South Africa; Lauren Stuart, Dr., Principal Investigator — WITS Health Hubb
Locations (4):
- Syddansk Universitet, Research Unit for Active Living, Department of Sports Science and Clinical Biomechanics, Odense, Denmark
- Amsterdam UMC, location Vrije Universiteit Amsterdam, Public and Occupational Health, Amsterdam, Netherlands
- Redeemer's University, Department of Physiotherapy, Osogbo, Nigeria
- University of the Witwatersrand, SAMRC Developmental Pathways for Health Research Unit, Faculty of Health Sciences, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
YoPA uses the approach "as open as possible, as restricted as necessary" as the leading principle in providing open access to research data, which includes taking measures to make research data findable, accessible, interoperable and reusable.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from July 2024.
Access Criteria: Only anonimized data will be shared as well as additional supporting information, like a co-creation protocol, data dictionary code book, topic lists for focus groups and interviews, etc. All results will be integrated in an open access YoPA toolbox targeted at academic researchers, public health practitioners and authorities, policy makers, and citizens.
  To request for data, a completed YoPA form "I want to reqest access to the YoPA data" should be submitted. Up to ten days after submission, the proposal will be evaluated by three members of the YoPA consortium.
  Please check for more information the YoPA website: https://www.yopa-project.eu/
URL: https://osf.io/rgkvu/

REFERENCES:
- [Background] Chinapaw MJM, Klaufus LH, Oyeyemi AL, Draper C, Palmeira AL, Silva MN, Van Belle S, Pawlowski CS, Schipperijn J, Altenburg TM. Youth-centred participatory action approach towards co-created implementation of socially and physically activating environmental interventions in Africa and Europe: the YoPA project study protocol. BMJ Open. 2024 Feb 21;14(2):e084657. doi: 10.1136/bmjopen-2024-084657. PMID 38387985
- See also: Related Info — https://doi.org/10.1136/bmjopen-2024-084657